CLINICAL TRIAL: NCT03428438
Title: Initial Education for Rehabilitation and Motivation Program Following a Myocardial Infarction. Rehabilitation Exercises at Home Via SMS or in the Hospital Physiotherapy Department
Brief Title: Initial Education for Rehabilitation and Motivation Program Following a Myocardial Infarction Via SMS or Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HYMC-0131-17
Record Dates: First submitted 2018-01-29; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-01

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Subjects recruited will be randomized into two groups: one group of subjects (the study group) A physical reminder by a physiotherapist, and a daily reminder of physical exercise by SMS on weekdays A through E. The second group (the control group) will be given a routine training in the ward by a nurse and you will receive a weekly SMS message
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group SMS to home phone (Other): A physical reminder by a physiotherapist, and a daily reminder of physical exercise by SMS on weekdays A through E.
  Interventions: Other: Rehabilitation at home via SMS
- Controlled group hospital based (Other): Physical rehabilitation in the ward physiotherapist
  Interventions: Other: Rehabilitation at home via SMS

INTERVENTIONS:
Other: Rehabilitation at home via SMS — Cardiac rehabilitation
  Other Names: Rehabilitation in hospital setting

SUMMARY:
The innovation in this preliminary study is the use of message reminders in patients after myocardial infarction in stage I of rehabilitation (ie discharge from hospital) at home via SMS, compared with studies of patients undergoing cardiac rehabilitation (stage II)in the hospital physiotherapy department.

DETAILED DESCRIPTION:
The first stage of rehabilitation begins during hospitalization. Motivation for the rehabilitation process for the patient. At this stage there will be preparation for release and guidance for the patient and their families regarding secondary prevention and return to domestic activity. This stage includes mobility, walking, controlled motility and gradual joint activation to maintain ranges and prevent complications from prolonged immobilization in bed.

ELIGIBILITY:
Inclusion Criteria:

Informed consent Criteria for inclusion Patients after acute myocardial infarction admitted to the intensive care unit Patients who speak the Hebrew language Patients with a cell phone to receive a reminder using a message

Exclusion criteria:

Orthopedic or neurological problem that would prevent physical activity. A score lower than 24 in the MoCA test. High-risk patients.

Complications: of myocardial infarction congestive heart failure, cardiogenic shock and / or ventricular arrhythmias.

Angina or shortness of breath at rest. Decrease >1mm in the ST segment in the ECG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac rehabilitation | 1 month
  Cardiac rehabilitation following heart attack following discharge

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Shotan, Prof, Principal Investigator — Hillel yaffe MC